CLINICAL TRIAL: NCT02826954
Title: The Nasal Airway in Chronic Obstructive Pulmonary Disease
Acronym: COPD
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2017
Record Dates: First submitted 2016-05-25; First posted 2016-07-11 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Paranasal Sinus Diseases; Nasal Obstruction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Paranasal Sinus Diseases; Nasal Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Nasal airway epithelial cells will be collected by the use of a nasal brush, and stored in a biobank.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients: Self administered questionnaires regarding sinonasal and lung symptoms, quality of life as well as symptoms of depression and anxiety.
  Lower airway assessment using Spirometry with reversibility Upper airway assessment using Acoustic Rhinometry, Rhinomanometry and Peak nasal Inspiratory Flow Nasal biopsy using a nasal brush Nasal endoscopy Allergic prick-test
  Interventions: Other: Upper airway assessment, including nasal biopsy
- Healthy subjects: Self administered questionnaires regarding sinonasal and lung symptoms, quality of life as well as symptoms of depression and anxiety.
  Lower airway assessment using Spirometry with reversibility Upper airway assessment using Acoustic Rhinometry, Rhinomanometry and Peak nasal Inspiratory Flow Nasal biopsy using a nasal brush Nasal endoscopy Allergic prick-test
  Interventions: Other: Upper airway assessment, including nasal biopsy

INTERVENTIONS:
Other: Upper airway assessment, including nasal biopsy

SUMMARY:
The study is based on the theory of a "unified airway" that considers the nose and paranasal sinuses together with lower airways as one integrated unit. The upper and lower respiratory tracts function as an interdependent physiologic mechanism, and stimuli that trigger changes in one portion of the airway, can provoke similar changes throughout the airway. This is well documented in asthmatic patients but documented poorly in patients suffering from chronic obstructive lung disease (COPD).

COPD is associated with sinonasal symptoms and decreased quality of life. Although nasal involvement has been found to directly affect the lower airway, sinonasal disease is under-diagnosed and under-treated in patients with COPD. This study is embedded in a larger project where the goal is to gain knowledge supporting the theory of a "unified airway" in patients with COPD.

Here sinonasal, pulmonary and generic health related quality of life will be studied in a group of patients with COPD versus a control group. The severity of nasal airway obstruction will be linked to the the severity of pulmonary airway obstruction. Assessment of pathological changes in the nose with nasal endoscopy, as well as performing a nasal cytological brushing for the identification of nasal inflammatory responses in the nose, will be conducted in both the control and study group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD: all stages
* Healthy individuals for the control group

Exclusion Criteria both groups:

* asthma
* systemic disease such as Cystic Fibrosis, Kartagener syndrome, sarcoidosis
* upper airway infection during the last 2 weeks
* COPD exacerbation during the last 6 weeks
* previous surgery in the nose and paranasal sinuses
* ongoing treatment for malignant disease
* severe depression, Alzheimers disease and Parkinson's disease
* pregnancy or nursing

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with chronic obstructive pulmonary disease (COPD) in St Olavs Hospital, Trondheim, Norway, and healthy participants matched in age and sex.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
pathological changes in the nose assessed with nasal endoscopy | 4 hours
inflammatory responses in the nose identified by nasal cytological brushing | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Wenche Thorstensen, PhD MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
Biobank 1